CLINICAL TRIAL: NCT06424613
Title: Investigating the Effects of Lithium Carbonate on Suicide and Self-harm in Adolescents and Young Adults With Bipolar Disorder in China
Brief Title: Effects of Lithium on Suicide Prevention in Adolescents and Young Adults With Bipolar Disorder in China
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: F2023-12-20-4-1
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Bipolar Disorder; Suicidal Ideation; Suicide, Attempted; Nonsuicidal Self Injury
Keywords: Lithium; Bipolar disorder; Suicide; Nonsuicidal Self Injury
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation; Suicide, Attempted; Self-Injurious Behavior; Suicide | interventions — Lithium Carbonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lithium Group
  Interventions: Drug: Lithium Carbonate
- Non-lithium Group
  Interventions: Drug: Non-lithium medication

INTERVENTIONS:
Drug: Lithium Carbonate — Participants must have been prescribed lithium for the past year and demonstrate at least 80% adherence to their lithium medication regimen during the first six months of the study period.
  Groups: Lithium Group
Drug: Non-lithium medication — No history of lithium use within the past year
  Groups: Non-lithium Group

SUMMARY:
This study aims to use a retrospective cohort approach to explore the impact of lithium carbonate on suicide and self-harm related events among adolescents and young adults with bipolar disorder in China.The primary objective of this study is to investigate the effects of lithium carbonate on suicidal ideation in adolescents and young adults with bipolar disorder in China. Secondary objectives include exploring its effects on preventing suicide attempts, non-suicidal self-injury, and aggressive behaviors in this population.

ELIGIBILITY:
Inclusion Criteria:

-

1 For Lithium group

1. Aged 12-45 years (adolescents 12-17, young adults 18-45).
2. Diagnosed with bipolar disorder using the the Mini-International Neuropsychiatric Interview (M.I.N.I.) (M.I.N.I.; version 5.0) based on Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria.
3. Adolescents diagnosed using the M.I.N.I. Kid version.
4. Lithium medication adherence of at least 80% in the first six months over the past year.
5. Not in an acute phase of illness.
6. Patient or guardian able to participate in assessment interviews.
7. Informed consent signed by participants and guardians (for adolescents).

2 for Non-lithium group

1. Aged 12-45 years (adolescents 12-17, young adults 18-45).
2. Diagnosed with bipolar disorder using the Mini-International Neuropsychiatric Interview (M.I.N.I.; version 5.0) based on DSM-IV criteria.
3. Adolescents diagnosed using the M.I.N.I. Kid version.
4. No lithium use over the past year.
5. Not in an acute phase of illness.
6. Patient or guardian able to participate in assessment interviews.
7. Informed consent signed by participants and guardians (for adolescents).

Exclusion Criteria:

1. Severe physical illness or active substance abuse.
2. Severe cognitive impairments, including developmental delays or dementia.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with bipolar disorder ranged in age from 12 to 45 years
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation | over the past year
  Measured using the Columbia Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Suicidal attempt | over the past year
  measured using the Columbia Suicide Severity Rating Scale (C-SSRS)
Non-suicidal self-injury | over the past year
Violent and aggressive behaviors | over the past year
  measured using the Chinese version of the Buss & Perry Aggression Questionnaire

OTHER OUTCOMES:
Depressive symptoms | over the past two weeks
  measured by Beck Depression Inventory
Mood symptoms | over the past year
  measured by Mood Disorder Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No